CLINICAL TRIAL: NCT03817866
Title: Chromogranin A as Surveillance Biomarker in Patients With cARcinoids (The CASPAR Study)
Brief Title: Chromogranin A as Blood Marker in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Brahms AG (Industry)
Responsible Party: Sponsor
Other Study IDs: Brahms-CASPAR
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Gastric Neoplasms; Pancreatic Neoplasms; Small Intestinal Neoplasms; Colorectal Neoplasms
Keywords: Endocrine tumors; Carcinoids; Functional NETs; Non-functional NETs; Immunoassay
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Carcinoid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BRAHMS CgA II KRYPTOR: Adult patients with well defined grade 1 and grade 2 GEP-NETs. Serial serum samples from all patients will be analyzed using the BRAHMS CgA II KRYPTOR Assay.
  Interventions: Diagnostic Test: BRAHMS CgA II KRYPTOR

INTERVENTIONS:
Diagnostic Test: BRAHMS CgA II KRYPTOR — The BRAHMS CgA II KRYPTOR kit is an automated immunofluorescent assay for the quantitative determination of the concentration of CgA in human serum.
  The assay is to be used as an aid in monitoring disease progression during the course of disease and treatment in patients with GEP-NETs (grade 1 and grade 2).
  Serial testing for patient BRAHMS CgA II KRYPTOR assay values should be used in conjunction with other clinical methods for monitoring GEP-NETs (grade 1 and grade 2).

SUMMARY:
Gastroentero-pancreatic neuroendocrine tumors (GEP-NETs) are a heterogenous group of neoplasms that arise from enterochromaffin cells of the gastrointestinal (GI) tract and pancreas. They account for 50-70% of all incident NETs. Due to the lack of symptoms in the early stage of disease and the frequency of nonspecific GI symptoms, GEP-NETs are difficult to diagnose.

Identification of effective biomarkers (such as Chromogranin A) to improve GEP-NET diagnosis, as well as to assess treatment efficacy, relapse and prognosis, is important for improving outcomes for patients with GEP-NETs.

The purpose of this study is to validate the performance of Brahms (BRAHMS) Chromogranin A II Kryptor (KRYPTOR) assay to monitor the course of disease in patients with well-defined GEP-NETs.

DETAILED DESCRIPTION:
A general characteristic for neuroendocrine tumors (NET) is expression of chromogranin A (CgA), which is released from neuroendocrine cells, occasionally together with cell specific hormones such as gastrin, insulin, somatostatin, and serotonin in functional tumors. Human CgA is an acidic 439 amino acid protein with a sequence containing several mono- and dibasic cleavage sites, and correspondingly, numerous fragments of CgA have been identified in tissue and plasma. CgA is critical to the formation of secretory granules that characterize NETs, and is therefore a useful marker for NETs.

Plasma concentrations of CgA and/or CgA fragments are elevated in most NETs. Moreover, since plasma CgA concentrations seem to be closely related to tumor burden in humans, plasma CgA concentration is an important prognostic factor. As such, high plasma concentrations of CgA as well as a dramatic increase in plasma CgA within a short time period, is associated with a poorer prognosis. Plasma CgA has also been suggested to be useful in the follow-up of patients with NETs.

Taken together, these observations support the notion that CgA is a promising biomarker candidate for monitoring treatment effectiveness and disease progression or regression.

Participation in this clinical study requires no additional visits to the oncologist, radiology or the laboratory. All information needed for the study will be obtained during typical visits as recommended by the oncologist. Clinical assessment of patients with GEP-NETs (according to NCCN guidelines) is based on physical exam, imaging (CT or MRI scans) and laboratory parameters. The course of disease is followed by RECIST 1.1 categorization including the evaluation of tumor burden by imaging.

ELIGIBILITY:
Inclusion Criteria:

* Primary well-differentiated G1 and G2 neuroendocrine tumor located in jejunum, ileum, colon, rectum, duodenum, appendix, stomach, or pancreas
* Measurable disease according to RECIST criteria (Version 1.1)
* Eighteen years of age or older
* CT or MRI order obtained and within 4 weeks of CgA measurement
* BRAHMS CgA II KRYPTOR baseline measurement available
* Patient has discontinued the following treatments for at least 3 weeks before study start: i) proton pump Inhibitors (PPI), ii) corticoids, iii) H2-receptor antagonists
* Baseline Eastern Cooperative Oncology Group Performance Scale (ECOG PS) <2
* Written informed consent signed

Exclusion Criteria:

* Other active malignancy with the exclusion of melanoma or other cancers that occurred more than 5 years ago
* Participation in another clinical trial involving an investigational therapeutic (exception: diagnostic studies and studies evaluating known therapies)
* No measurable disease by RECIST criteria (Version 1.1)
* Severe renal dysfunction defined as creatinine of 1.5x upper limit of normal (ULN)
* Severe liver dysfunction in the absence of liver metastasis defined by aspartate aminotransferase (AST), serum total bilirubin and/or alanine transaminase (ALT) 1.5x ULN; severe liver dysfunction in the presence of liver metastasis defined by AST and ALT over 5x ULN and total bilirubin over 1.5x ULN
* Severe gastrointestinal disorders (chronic atrophic gastritis, pancreatitis, inflammatory bowel disease, irritable bowel syndrome)
* Severe cardiovascular disease (severe symptomatic congestive heart failure, pulmonary artery hypertension, acute coronary syndrome)
* Patients receiving active treatment with the following medications and samples were collected less than 3 weeks after discontinuing: i) proton pump Inhibitors (PPI), ii) corticoids, iii) H2-receptor antagonists
* Chronic alcohol and/or substance abuse
* Known pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with diagnosed well-differentiated G1 and G2 GEP-NETs
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Disease Progression | 36 months
  Progression vs. non-progression in patients with well-defined GEP-NETs assessed by RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Halperin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (3):
  - Stanford University Medical Center, Palo Alto, California
  - Mayo Clinic, Rochester, Minnesota
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- See also: National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines — https://www.nccn.org/professionals/physician_gls/default.aspx